CLINICAL TRIAL: NCT02523755
Title: Evaluation of Regional Distribution of Ventilation in Spontaneous Breathing Patients During Labor With or Without Epidural Analgesia Using EIT (Electrical Impedance Tomography)
Brief Title: Evaluation of Regional Distribution of Ventilation During Labor With or Without Epidural Analgesia
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Universitair Ziekenhuis Brussel (Other)
Responsible Party: Principal Investigator, Veerle Van Mossevelde, Data Nurse, Universitair Ziekenhuis Brussel
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: EIT
Record Dates: First submitted 2015-07-28; First posted 2015-08-14 (Estimated); Last update posted 2016-12-06 (Estimated); Status verified 2016-12

CONDITIONS: Pregnancy; Atelectasis
Keywords: epidural analgesia for labor; respiratory function; electrical impedance tomography
MeSH Terms: conditions — Pulmonary Atelectasis; Respiratory Aspiration

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Epidural analgesia Ropivacaine (Active Comparator): Placement of an epidural catheter to achieve pain relief
  Interventions: Drug: Epidural analgesia Ropivacaine; Drug: Absence of epidural analgesia
- Absence of epidural analgesia (Sham Comparator): No placement of an epidural catheter either because of patient refusal or contraindication
  Interventions: Drug: Epidural analgesia Ropivacaine; Drug: Absence of epidural analgesia

INTERVENTIONS:
Drug: Epidural analgesia Ropivacaine — Measurement of regional distribution as assessed by EIT before and after injection of local anesthetics
Drug: Absence of epidural analgesia — Measurement of regional distribution as assessed by EIT before and after delivery

SUMMARY:
With an efficient epidural analgesia the physiological effects of pain are disabled during labor. Pain may cause an increase of minute volume, oxygen consumption and a decrease of paCO2 (Arterial CO2 pressure). The study will evaluate the lung function before and after labor with and without epidural analgesia. With more efficient breathing, the occurence of atelectasis should be reduced; this effect will be investigated in these settings for the first time with the electrical impedance tomography, which is a completely non-invasive measure.

DETAILED DESCRIPTION:
The bedside efficacy of the electrical impedance tomography (EIT) in intensive care settings during mechanical ventilation is known. However, no studies demonstrate its utility during epidural analgesia for labor.

The purpose of this study is to evaluate lung function and atelectasis in pregnant women with or without epidural analgesia, during labor and after delivery.

Only adult consenting patients ASA I & ASA II (American Society of Anaesthesiologists) are included in the study. According to institutional protocols lumbal epidural catheter is inserted and tested at the start of the labor, while patients' parameters are monitored.

Refusal to epidural analgesia, technical difficulties to insert the epidural catheter or any medical contraindication will result in inclusion of these patients in the control group.

Measurement with EIT is not invasive and harmful neither for the mother nor for the child.

It consists of putting a belt around the chest; this belt is linked to a monitor which measures the impedance of the different lung regions.

Electrical impedance measurements will be done for short periods of maximum 5 min. each as follows:

1. Placement before injection of local anesthetics through the epidural catheter in the study goup; in the control subset placement of the belt will be done when an epidural anesthetic would have been considered.
2. 1 hour after placement of the belt
3. 1 hour after delivery

These periods will be compared.

ELIGIBILITY:
Inclusion Criteria:

* ASA I
* ASA II

Exclusion Criteria:

* Caesarian
* < 18 years
* Expulsions

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2015-09; Primary Completion 2016-11 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Better lung function after labor with epidural analgesia | 24h
  Using EIT we will map the degree of atelectasis

CONTACTS AND LOCATIONS:
Overall Officials: Maxim Doutreluigne, MD, Principal Investigator — Universitair Ziekenhuis Brussel; Laszlo L Szegedi, Prof., Study Chair — Universitair Ziekenhuis Brussel
Locations (1):
- Universitair Ziekenhuis Brussel, Jette, Vlaams Brabant, Belgium

IPD SHARING:
Plan to Share IPD: No